CLINICAL TRIAL: NCT00330434
Title: Human CYP2B6: Induction by Ethanol and Polymorphisms
Brief Title: Effect of Ethanol and Genetic Polymorphisms on Bupropion Metabolism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was a F32 Fellowship. Trial was proposed however Principle Investigator does not believe trial took place.
Sponsor: Tufts University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAGRE15647; F32AA015647-01A1 (NIH); 1F32AA015647-01A1 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Drinking; Depression; Smoking Cessation; Attention Deficit Disorder
Keywords: Alcohol; Bupropion; Chlorzoxazone; Interaction; Induction; Depression; Smoking; Drinking; Cytochrome P450 Enzyme; CYP2B6; CYP2E1; Pharmacogenetics; Pharmacokinetics; Pharmacodynamics; Boston; Tufts University
MeSH Terms: conditions — Alcohol Drinking; Depression; Smoking Cessation; Attention Deficit Disorder with Hyperactivity; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial Withdrawn 2 (Other): Trial Withdrawn 2
  Interventions: Other: Trial Withdrawn 2
- Trial Withdrawn 1 (Other): Trial Withdrawn 1
  Interventions: Other: Trial Withdrawn 1

INTERVENTIONS:
Other: Trial Withdrawn 1 — Trial Withdrawn 1
  Arms: Trial Withdrawn 1
Other: Trial Withdrawn 2 — Trial Withdrawn 2
  Arms: Trial Withdrawn 2

SUMMARY:
The two purposes of this study are

1. to determine what effect the chronic and moderate/heavy drinking of alcoholic beverages has

   1. on the blood level of bupropion and chlorzoxazone and their major breakdown products in the blood and
   2. on the stimulant effect of bupropion and
2. to determine what effect a normal and common (25% frequency) genetic variation of a specific liver enzyme (that breaks down bupropion) has

   1. on the blood levels of bupropion and its major breakdown products in the blood and
   2. on the stimulant effect of bupropion.

Two groups of volunteers will be recruited for this study:

1. volunteers who drink moderate to heavy amounts of alcohol frequently and
2. volunteers who usually do not drink alcohol.

Volunteers will NOT be asked to change their drinking (or nondrinking) habits during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are 21 - 55 years of age.
* Either 1) Moderate-to-heavy drinkers who drink on average more than 14 but less than 28 drinks per week; OR 2) adults who normally abstain from drinking alcohol.

Exclusion Criteria:

* Participants who are currently taking prescription medications (including oral contraceptives)
* Pregnancy
* Body mass index (BMI) greater than 30
* History of seizures or eating disorders

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Greenblatt, MD, Principal Investigator — Tufts University; Chair of Department of Pharmacology and Experimental Therapeutics, Sackler School; Michael H. Court, BVsc, PhD, Principal Investigator — Tufts University, Department of Pharmacology and Experimental Therapeutics, Sackler School
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hesse LM, Venkatakrishnan K, Court MH, von Moltke LL, Duan SX, Shader RI, Greenblatt DJ. CYP2B6 mediates the in vitro hydroxylation of bupropion: potential drug interactions with other antidepressants. Drug Metab Dispos. 2000 Oct;28(10):1176-83. PMID 10997936
- [Background] Hesse LM, He P, Krishnaswamy S, Hao Q, Hogan K, von Moltke LL, Greenblatt DJ, Court MH. Pharmacogenetic determinants of interindividual variability in bupropion hydroxylation by cytochrome P450 2B6 in human liver microsomes. Pharmacogenetics. 2004 Apr;14(4):225-38. doi: 10.1097/00008571-200404000-00002. PMID 15083067